# STATISTICAL ANALYSIS PLAN PHASE II-III

**VERSION:** 

2.0

**STUDY DRUG:** 

<sup>18</sup>F-DCFPyL Injection (PyL)

**PROTOCOL** 

NUMBER: PyL-2301

NCT02981368

## **STUDY TITLE:**

A Pr**O**spective Phase 2/3 Multi-Center **S**tudy of <sup>18</sup>F-DCF**P**yL PET/CT Imaging in Subjects with P**R**ostate Cancer: **E**xamination of Diagnostic Accurac**Y** (OSPREY)

#### **SPONSOR:**

Progenics Pharmaceuticals, Inc.
One World Trade Center
47<sup>th</sup> Floor, Suite J
New York, NY 10007
646-975-2500

This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

# **SIGNATURE PAGE**



# TABLE OF CONTENTS

| 1. | LIST OF ABBREVIATIONS | 8 |
|---|---|---|
| 2. | INTRODUCTION | 11 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 12 |
| 3.1. | Study Objectives | 12 |
| 3.1.1. | Primary Objective | 12 |
| 3.1.2. | Secondary Objectives | 12 |
| 3.1.3. | Exploratory Objectives | 12 |
| 3.2. | Efficacy Endpoints | 12 |
| 3.2.1. | Primary Efficacy Endpoints | 12 |
| 3.2.2 | Secondary Efficacy Endpoints | 13 |
| 3.2.3 | Exploratory Efficacy Endpoints | 13 |
| 3.3. | Safety Endpoints | 13 |
| 4. | STUDY DESIGN | 14 |
| 4.1. | Summary of Study Design | 14 |
| 4.2. | Definition of Study Drugs and Treatment Follow-up | 14 |
| 4.3. | Sample Size | 15 |
| 4.4. | Randomization | 16 |
| 4.5. | Clinical Assessments | 16 |
| 4.6. | Interim Analyses | 17 |
| 4.7. | Final Analyses | 17 |
| 5. | GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING | 18 |
| 5.1. | General Summary Table and Individual Subject Data Listing Considerations | 18 |
| 5.2. | General Post Text Summary Table and Individual Subject Data Listing Format Considerations | 18 |
| 5.3. | Data Presentation Conventions | 18 |
| 5.4. | Analysis Populations | 18 |
| 5.4.1. | Consented Set | 18 |
| 5.4.2. | Safety Set | 18 |
| 5.4.3. | Evaluable Set | 19 |
| 5.4.4. | Change in Planned Protocol Procedure Set | 19 |
| 5 4 5 | Per Protocol Set | 19 |

| $\mathcal{C}$ | s Pharmaceuticals, Inc.<br>l Analysis Plan – Protocol PyL-2301 | September 5, 2018 |
|---|---|---|
| 5.4.6. | PK Blood Set | 19 |
| 5.4.7. | PK Urine Set | 19 |
| 5.5. | Derived and Transformed Data | 19 |
| 5.5.1. | Baseline Definition | 19 |
| 5.5.2. | Baseline Age | 19 |
| 5.5.3. | Study Day | 19 |
| 5.5.4. | Change and Percent Change from Baseline | 19 |
| 5.5.5. | Prior and Concomitant Medications | 20 |
| 5.5.6. | Treatment-Emergent Adverse Events | 20 |
| 5.5.7. | Sensitivity, Specificity, PPV, and NPV | 20 |
| 5.5.8. | Lesions Per Subject | 24 |
| 5.5.9. | Visit Windows | 25 |
| 5.5.10. | Decay Corrected Dose at Time of Administration | 25 |
| 5.5.11. | Lesion location defined from SUV values | 25 |
| 5.5.12. | Change in Clinical Management Plan from Questionnaire | 26 |
| 5.5.13. | PSA groups | 26 |
| 5.5.14. | Gleason Scores | 26 |
| 5.5.15. | Prior Prostate Cancer History and Therapies | 27 |
| 5.5.16. | Estimate GFR. | 27 |
| 5.5.17. | Renal impairment | 27 |
| 5.5.18. | Laboratory Parameter Unit Conversions | 28 |
| 5.6. | Handling of Missing Data | 29 |
| 5.6.1. | Missing Efficacy Endpoints | 29 |
| 5.6.2. | Missing Start and Stop Dates for Concomitant Medication | 29 |
| 6. | STUDY POPULATION | 31 |
| 6.1. | Disposition | 31 |
| 6.2. | Protocol Deviations | 31 |
| 6.3. | Demographic and Baseline Characteristics | 31 |
| 6.4. | Medical History, including Prostate Cancer History | 31 |
| 6.5. | Prior Prostate Cancer Therapies and Surgeries | 31 |
| 6.6. | Prior Medication History and Medications Present at Entry | 32 |
| 6.7. | Conventional Imaging at Baseline | 32 |
| 7. | EFFICACY | 32 |

| _ | es Pharmaceuticals, Inc. al Analysis Plan – Protocol PyL-2301 Se | ptember 5, 2018 |
|---|---|---|
| 7.1. | General Considerations. | 32 |
| 7.2. | Testing Statistical Assumptions Including Comparability at Baseline. | 32 |
| 7.2.1. | Test of Proportions | 32 |
| 7.2.2. | Test of means | 32 |
| 7.3. | Statement of the Null and Alternate Hypotheses | 33 |
| 7.4. | Subgroup Analyses | 33 |
| 7.5. | Multiple Comparisons and Multiplicity | 33 |
| 7.6. | Analysis of the Primary Efficacy Endpoint | 33 |
| 7.6.1. | Primary Efficacy Analysis of Primary Endpoints | 33 |
| 7.6.2. | Sensitivity Analyses of the Primary Endpoints | 33 |
| 7.7. | Analysis of Secondary Efficacy Endpoints | 34 |
| 7.7.1. | NPV and PPV in Cohort A | 34 |
| 7.7.2. | PPV and Sensitivity in Cohort B | 34 |
| 7.7.3. | Detection Rates for Lesion Counts in both Cohorts Combined | 34 |
| 7.7.4. | PK | 34 |
| 7.8. | Analysis of Exploratory Endpoints | 35 |
| 7.9. | Reader Reliability | 36 |
| 7.9.1. | Intra-Reader Reliability | 36 |
| 7.9.2. | Inter-Reader Reliability | 36 |
| 8. | SAFETY AND TOLERABILITY | 37 |
| 8.1. | Adverse Event Preferred Term and System Organ Class Summary Ta | bles37 |
| 8.1.1. | Summaries of Adverse Event Incidence Rates for All Subjects | 37 |
| 8.1.2. | Summaries of Adverse Incidence Rates for Serious Adverse Events (State Adverse Event Discontinuations, and Death | |
| 8.2. | Exposure to Study Drug | 38 |
| 8.3. | Concomitant and Other Medications | 38 |
| 8.4. | Routine Laboratory Data | 38 |
| 8.5. | Vital Signs | 38 |

8.6.

8.7.9.

9.1.

| _ | cs Pharmaceuticals, Inc.<br>cal Analysis Plan – Protocol PyL-2301 | September 5, 2018 |
|---|---|---|
| 10. | PLANNED TREATMENT SAP CHANGES THA PROTOCOL | |
| 11. | REFERENCES | 41 |
| 12. | APPENDIX | 43 |
| 12.1. | Table of Contents for Data Display Specifications | 43 |

| Progenics | Pharmaceutic | eals, Inc. | |
|-------------|---------------|--------------|----------|
| Statistical | Analysis Plai | n – Protocol | PyL-2301 |

September 5, 2018

# LIST OF TABLES

| Table 1: | List of Abbreviations | 8 |
|---|---|---|
| Table 2: | Schedule of Assessments | 16 |
| Table 3: | Classification of <sup>18</sup> F-DCFPyL Imaging Result and Histopathology Result | 20 |
| Table 4: | List of Tables, Listings and Figures | 43 |
| | LIST OF FIGURES | |
| Figure 1: | Study Schema | 15 |

# 1. LIST OF ABBREVIATIONS

**Table 1: List of Abbreviations** 

| Abbreviation | Term |
|---|---|
| <sup>18</sup> F | fluorine 18 |
| ADT | androgen deprivation therapy |
| AE | adverse event |
| ATC | anatomical therapeutic classification |
| AUC | area under the curve |
| BN | bone |
| BP | blood pressure |
| CI | confidence interval |
| C <sub>max</sub> | maximum observed concentration |
| CL | clearance |
| cm | centimeter |
| СРМ | counts per minute |
| CT | computed tomography |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| eGFR | estimated Glomerular filtration rate |
| ePLND | Extended lymph node dissection in prostate cancer |
| FN | false negative |
| FP | false positive |
| HR | heart rate |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| I(p) | total positive imaging |
| I(n) | total negative imaging |
| Kg/m <sup>2</sup> | kilograms per metered squared |
| LLN | lower limit of normal |
| LN | lymph node |
| MBq | Megabecquerel |
| mCi | millicurie |
| MDRD | Modification of diet in renal disease study |

**Table 1: List of Abbreviations** 

| Abbreviation | Term |
|---|---|
| MedDRA | Medical Dictionary for Regulatory Activities |
| mL | milliliter |
| MRI | magnetic resonance imaging |
| MRT | mean residence time |
| NC | North Carolina |
| ng/mL | nanogram/milliliter |
| NPV | negative predictive value |
| PET/CT | positron emission tomography/computed tomography |
| PK | pharmacokinetics |
| PPV | positive predictive value |
| PSA | prostate specific antigen |
| PSMA | Prostate specific membrane antigen |
| PT | preferred term |
| R(n) | total negative histopathology |
| R(p) | total positive histopathology |
| RP | radical prostatectomy |
| RR | respiratory rate |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SCr | serum creatinine |
| SD | standard deviation |
| SOC | system organ class |
| ST | Soft tissue |
| SUV <sub>max</sub> | maximum standardized uptake value |
| SUV <sub>mean</sub> | Mean standardized update value |
| $SUV_{peak}$ | peak standardized uptake value |
| $SUV_r$ | ratio to reference tissue standardized uptake value |
| TEAE | treatment-emergent adverse event |
| T <sub>1/2</sub> | half life |
| T <sub>1/2alpha</sub> | alpha phase distributive half life |
| T <sub>1/2beta</sub> | beta phase elimination help life |

**Table 1: List of Abbreviations** 

| Abbreviation | Term |
|----------------------|-------------------------------------------|
| T <sub>1/2elim</sub> | elimination half life |
| $T_{\text{max}}$ | time to maximum concentration |
| TN | true negative |
| TOA | time of administration |
| TP | true positive |
| ULN | Upper limit of normal |
| USA | United States of America |
| $V_{ss}$ | steady state volume of distribution |
| WHODD | World Health Organization Drug Dictionary |

#### 2. INTRODUCTION

The statistical analysis plan (SAP) is based on:

- Protocol amendment 2 dated November 6, 2017,
- ICH guidelines E6<sup>1</sup> and E9<sup>2</sup>.

The purpose of this document is to provide details about study populations, how variables will be derived, how missing data will be handled as well as details about statistical methods to be used to analyze the safety and efficacy data from Study PyL-2301.

The list of tables, listings and their shells are guidelines which may be refined to facilitate programming. Such changes will not be documented in an amendment to this document. However, any changes to populations, endpoints or analysis methods will be documented in a SAP amendment and will be noted in the clinical study report, as relevant.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

## 3.1. Study Objectives

#### 3.1.1. Primary Objective

The primary objective of the study is to assess the diagnostic performance of <sup>18</sup>F-DCFPyL PET/CT imaging to determine the presence or absence of metastatic disease in pre-prostatectomy subjects with high risk prostate cancer (cohort A).

#### 3.1.2. Secondary Objectives

- 1. To evaluate the safety and tolerability of <sup>18</sup>F-DCFPyL
- 2. To assess the diagnostic performance of <sup>18</sup>F-DCFPyL PET/CT imaging to determine the presence or absence of prostate cancer within sites of metastasis or local recurrence (cohort B).
- 3. To determine detection rates of <sup>18</sup>F-DCFPyL PET/CT and conventional imaging among lesion locations (e.g., bone, lymph nodes, soft tissue, prostate gland)
- 4. To determine positive and negative predictive value (PPV and NPV) of <sup>18</sup>F-DCFPyL PET/CT imaging
- 5. To determine the pharmacokinetics, bio-distribution and excretion of <sup>18</sup>F-DCFPyL

## 3.1.3. Exploratory Objectives

- 1. To assess <sup>18</sup>F-DCFPyL uptake among lesion locations (e.g., bone, lymph nodes, soft tissue, prostate gland)
- 2. To assess the relationship between <sup>18</sup>F-DCFPyL uptake in prostatic and extra-prostatic lesions with baseline PSA and testosterone levels and Gleason Score at time of radical prostatectomy
- 3. To assess the diagnostic performance of <sup>18</sup>F-DCFPyL PET/CT imaging to detect prostate cancer within the prostate gland (Cohort A)
- 4. To assess the impact of <sup>18</sup>F-DCFPyL PET/CT imaging on clinical management plan
- 5. To determine PPV of <sup>18</sup>F-DCFPyL PET/CT imaging for lesions detected by PET that are outside the planned surgical template or biopsy site

## 3.2. Efficacy Endpoints

#### 3.2.1. Primary Efficacy Endpoints

- 1. Specificity of <sup>18</sup>F-DCFPyL PET/CT imaging to determine the absence of metastatic prostate cancer within the pelvic lymph nodes relative to histopathology in Cohort A
- 2. Sensitivity of <sup>18</sup>F-DCFPyL PET/CT imaging to determine the presence of metastatic prostate cancer within the pelvic lymph nodes relative to histopathology in Cohort A

#### 3.2.2 Secondary Efficacy Endpoints

- 1. Sensitivity of <sup>18</sup>F-DCFPyL PET/CT imaging to detect prostate cancer within sites of metastasis or local recurrence relative to histopathology in Cohorts B
- 2. Comparison of detection rates for lesion counts overall and by location (i.e., bone, lymph nodes, soft tissue, prostate gland) between <sup>18</sup>F-DCFPyL PET/CT and conventional imaging in Cohorts A and B combined
- 3. PPV of <sup>18</sup>F-DCFPyL PET/CT imaging to predict prostate cancer within the prostate gland and lymph nodes in Cohort A
- 4. NPV of <sup>18</sup>F-DCFPyL PET/CT imaging to predict the absence of prostate cancer within the prostate gland and lymph nodes in Cohort A
- 5. PPV of <sup>18</sup>F-DCFPyL PET/CT imaging to predict prostate cancer within sites of local recurrence and other metastatic lesions in Cohort B
- 6. Pharmacokinetic parameters derived from blood samples [e.g., C<sub>max</sub>, area under the curve (AUC), total clearance (CL), steady-state volume of distribution (V<sub>ss</sub>), and mean residence time (MRT)] (subset of Cohorts A and B combined)

#### 3.2.3 Exploratory Efficacy Endpoints

- 1. <sup>18</sup>F-DCFPyL uptake in different lesion locations as defined by SUV<sub>peak</sub>, SUV<sub>max</sub>, and SUV<sub>r</sub> results derived from central readers for cohorts A and B combined and compared between histology outcomes
- 2. To assess the relationship between SUV<sub>peak</sub>, SUV<sub>max</sub>, volume, and SUVr and Gleason Score at time of radical prostatectomy, baseline PSA, and testosterone levels for both cohorts
- 3. Sensitivity of <sup>18</sup>F-DCFPyL PET/CT imaging within the prostate gland relative to histopathology in Cohort A
- 4. Specificity of <sup>18</sup>F-DCFPyL PET/CT imaging within the prostate gland relative to histopathology in Cohort A
- 5. Changes to clinical management based on a review of clinical and radiographic subject data before and after <sup>18</sup>F-DCFPyL PET/CT imaging by a central panel of disease experts using a structured questionnaire (Cohort A only)
- 6. PPV of <sup>18</sup>F-DCFPyL PET/CT imaging in subjects with corresponding histopathology for subjects who had a change in the planned protocol procedure (Both Cohorts combined)

## 3.3. Safety Endpoints

- 1. Treatment-emergent adverse events (TEAEs) and SAEs
- 2. Change from baseline in clinical laboratory parameters
- 3. Change from baseline in ECGs
- 4. Change from baseline in vital signs
- 5. Concomitant medication use

#### 4. STUDY DESIGN

## 4.1. Summary of Study Design

This is an open-label, non-randomized, Phase 2/3, multi-center study designed to evaluate the safety and diagnostic performance of <sup>18</sup>F-DCFPyL PET/CT imaging to determine the presence or absence of metastatic prostate cancer in subjects with high risk prostate cancer who were planned for radical prostatectomy with pelvic lymph node dissection (cohort A), and subjects with radiologic evidence of local recurrence or new or progressive metastatic disease (cohort B) who were biopsied if a positive lesion was found on the <sup>18</sup>F-DCFPyL PET/CT scan. The physician has the option to change the planned protocol specified procedure (i.e., RP ePLND for Cohort A subjects and Biopsy for Cohort B subjects) for the subjects based on the <sup>18</sup>F-DCFPyL PET/CT scan. The details of these changes will be collected on the CRF, and these subjects obviating the planned procedure will not be included in any of the primary or secondary endpoints.

Eligible subjects will be enrolled in a non-randomized, sequential manner, with competitive enrollment between study sites. Ten (10) study sites will be used in the U.S. and Canada.

Diagnostic performance characteristics of <sup>18</sup>F-DCFPyL PET/CT imaging will be evaluated using histopathology as the truth standard. Three independent readers from a central imaging core lab will be given access to <sup>18</sup>F-DCFPyL PET/CT imaging, conventional imaging, and biopsy-guided imaging. The central readers will be blinded to all other clinical information (i.e. pathology data) and radiology assessments. Likewise, local pathologists who generate the histopathology results for the primary endpoint are blinded to all imaging results.

A change in clinical management questionnaire will be filled out by an independent urologist who is not otherwise a participant of the study. To maintain the blind for imaging, a statistician who is independent from the PyL study team will generate subject listings. A combination of imaging and clinical data will then be posted to a share point site where the independent urologist will review these data and fill out the questionnaire based on the results he sees prior to PyL imaging and then again after PyL imaging. To keep things simple, only imaging data from reviewer 1 will be presented for this assessment to be performed.

## 4.2. Definition of Study Drugs and Treatment Follow-up

All subjects will be administered  $9 \pm 1$  mCi  $(333 \pm 37 \text{ MBq})^{18}\text{F-DCFPyL}$  injection followed by PET/CT imaging and either a biopsy or prostatectomy and lymphadenectomy as illustrated in the white boxes in Figure 1. These are the protocol's planned procedures. If a Physician decides to change these planned procedures after PET/CT imaging is obtained, subjects in Cohort A would not have surgery and subjects in Cohort B would not have a conventional imaging guided biopsy. These changes in planned protocol procedures are listed in the shaded boxes below. This should be a small number of subjects who will not be included in the primary analysis of the primary endpoint or any of the secondary endpoints.

Figure 1: Study Schema



If the subject did not want to go through with this planned procedure or withdrew from the study then this would not constitute a change in planned protocol procedure. If the planned procedure was intended but could not be completed, then this is also not a change in planned procedure.

## 4.3. Sample Size

The primary analysis in Cohort A will test the co-primary endpoints of sensitivity and specificity of <sup>18</sup>F-DCFPyL PET imaging relative to histopathology for the evaluable set of subjects in Cohort A with metastatic disease. For each co-primary endpoint, there will be three independent imaging readers. At least two of the three readers must reject the null hypothesis for specificity to be deemed a success. If specificity is a success, then the same two readers need to reject the null hypothesis for sensitivity leading to overall success of the primary endpoint. The null hypotheses will be tested in the following order:

- 1. Specificity of <sup>18</sup>F-DCFPyL PET imaging relative to histopathology in Cohort A  $H_0$ :  $\pi_{Sp} = 0.80$  versus  $H_1$ :  $\pi_{Sp} \neq 0.80$
- 2. Sensitivity of <sup>18</sup>F-DCFPyL PET/CT imaging relative to histopathology in Cohort A  $H_{01}$ :  $\pi_{Se} = 0.40$  versus  $H_{11}$ :  $\pi_{Se} \neq 0.40$

where  $\pi_{Se}$  is the true sensitivity and  $\pi_{Sp}$  is the true specificity of <sup>18</sup>F-DCFPyL PET imaging.

A total of 262 subjects from Cohort A will provide 80% power to reject the null hypothesis about sensitivity at the 5% significance level if the true sensitivity is at least 60% and at least 80% power to reject the null hypothesis about specificity at the 5% significance level if the true specificity is at least 87.8%. These calculations are based on the following assumptions:

• the probability of a positive histopathology sample in Cohort A is 20%,

The sample size is based on the normal approximation to the binomial distribution without a continuity correction<sup>3</sup>.

$$n \ge \left\{ \frac{z_{\alpha/2} \sqrt{P_0(1 - P_0)} + z_{\beta} \sqrt{P_1(1 - P_1)}}{P_1 - P_0} \right\}^2$$

where P<sub>0</sub> are P<sub>1</sub> are values of sensitivity under the null and alternative hypotheses, respectively. After adjusting sensitivity and specificity separately by their corresponding prevalence values, a total in 236 subjects are needed. Assuming a 10% drop out or non-evaluable rate increases the required number of subjects in Cohort A to 262.

The type I error rate will be preserved at 5% by requiring that both null hypotheses be rejected to draw the conclusion that <sup>18</sup>F-DCFPyL is efficacious for imaging. The second primary endpoint is only tested if the first primary endpoint is rejected at the 0.05 level of significance per a fixed sequential method. If the first hypothesis fails to be rejected, no further testing will be conducted.

No formal power calculations will be performed for Cohort B since it is not a primary endpoint. Approximately 115 subjects will be dosed in this cohort.

#### 4.4. Randomization

This study is not randomized. One treatment will be administered.

#### 4.5. Clinical Assessments

See Table 2 for the schedule of study assessments.

**Table 2: Schedule of Assessments** 

| | Screening/<br>Baseline | <sup>18</sup> F-DCFPyL<br>Dosing | <sup>18</sup> F-DCFPyL<br>Imaging | Pre-Surgery/<br>Biopsy<br>Follow-Up |
|---|---|---|---|---|
| | Day -30 to<br>Day 1 | Day 1 | 1-2 Hours<br>Post-Dosing | Within 28<br>Days Post-<br>Dosing |
| Cohorts A and B | | | | |
| Informed Consent & Eligibility | X | | | |
| Demographics (date of birth, race, ethnicity, height, weight) | X | | | |
| Medical History | X | | | |
| Prior Cancer Medications & Treatments | X | | | |
| Clinical Labs (hematology, chemistry) | X <sup>1</sup> | | | X |
| PSA (total) & Testosterone | X <sup>1</sup> | | | |
| Vital Signs (blood pressure, heart rate, temperature, respiratory rate) | X | X<br>(pre-dosing) | X (pre-imaging) | X |
| 12-Lead ECG | | X (pre-dosing) | X (pre-imaging) | |
| <sup>18</sup> F-DCFPyL Administration | | X | | |
| Whole Body PET/CT | | | X | |

**Table 2: Schedule of Assessments** 

| | Screening/<br>Baseline | <sup>18</sup> F-DCFPyL<br>Dosing | <sup>18</sup> F-DCFPyL<br>Imaging | Pre-Surgery/<br>Biopsy<br>Follow-Up |
|---|---|---|---|---|
| | Day -30 to<br>Day 1 | Day 1 | 1-2 Hours<br>Post-Dosing | Within 28<br>Days Post-<br>Dosing |
| Adverse Events | | 2 | X | X <sup>5</sup> |
| Concomitant Medications | X | X | | X |
| Conventional Imaging (CT or MRI, bone scan) | X <sup>2</sup> | | | |
| Surgery or Image-Guided Biopsy | | | | X <sup>3,6</sup> |
| Subset of Cohort A or B at Johns Hopkins Universi | Subset of Cohort A or B at Johns Hopkins University only for PK Analysis | | | |
| Blood Collection | | X <sup>4</sup> (9 collections) | | |
| Urine Collection | | X <sup>4</sup> (3 collections) | | |
| Whole Body PET/CT | | | X <sup>4</sup> (3 scans) | |

<sup>1</sup> To be collected prior to dosing, if collected on day of dosing. If PSA and testosterone have not been tested within 30 days of study drug injection, a blood draw will be collected prior to dosing.

- 3 Surgery or biopsy to occur at least 12 hours from time of <sup>18</sup>F-DCFPyL dosing but not more than 28 days from dosing. In Cohort B, imaging used to guide biopsy (i.e., CT, MRI) will be submitted to a central core imaging lab.
- 4 Analysis should occur immediately following last sample collected.
- 5 A safety phone call will also occur  $7(\pm 3)$  days post dosing [if surgery, biopsy or a change in planned protocol procedure has not yet occurred] and  $21(\pm 7)$  days post biopsy for just the subjects who had a conventional image guided biopsy in Cohort B.
- <sup>6</sup> If a subject's planned procedure (RP or biopsy) for prostate cancer changes following <sup>18</sup>F-DCFPyL imaging, the alternate or additional prostate cancer procedure and corresponding histopathology data will be recorded in the electronic case report form (eCRF).

#### 4.6. Interim Analyses

No interim analysis is planned for this study.

## 4.7. Final Analyses

The final analysis will be conducted after the database is locked.

<sup>2</sup> If not obtained as standard of care  $\leq$ 6 weeks (Cohort A) or  $\leq$  4 weeks (Cohort B) prior to Day 1. If Na- $^{18}$ F-PET bone scans conducted at screening must be at least 10 hours prior to dosing.

# 5. GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING

# 5.1. General Summary Table and Individual Subject Data Listing Considerations

Adverse event and medical history verbatim terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 4.0. Medications will be coded using the World Health Organization Drug Dictionary (WHODDE) from December 2016.

Summary tables and listings will include the following information: dataset(s) used in table production, date of data extract, date of output generation, the SAS program name and location (directory path), page x of y numbering. Adverse event and medical history summaries will indicate the MedDRA version; prior and concomitant medication summaries will indicate the WHODD version.

Summary tables for demographics and baseline characteristics, medical history, exposure, concomitant medications, and safety will include the following columns: Cohort A, Cohort B, overall (Cohorts A and B combined). Efficacy tables will be produced by cohort.

# 5.2. General Post Text Summary Table and Individual Subject Data Listing Format Considerations

Statistical analyses will be performed, and datasets and tables will be generated using SAS version 9.4 (SAS Institute, Inc., Cary, NC, USA).

#### 5.3. Data Presentation Conventions

Continuous data will be summarized using descriptive statistics [i.e., N, arithmetic mean, standard deviation (SD), median, minimum, and maximum]. The minimum and maximum will be displayed to the same level of precision as collected data; mean and median will be displayed to one level of precision greater than the data collected; SD will be displayed to two levels of precision greater than the data collected. Categorical data will be described using frequencies and percentages. A row for missing values will be included, when applicable. P-values will be presented at four decimal places.

Dates will be presented in DDMMMYY format and times will be presented as HH:MM using a 24-hour clock.

In tables and listings, columns of data will be decimal aligned.

## 5.4. Analysis Populations

#### **5.4.1.** Consented Set

All subjects who sign an informed consent document will be included in the consented set.

#### 5.4.2. Safety Set

All subjects who receive any amount of <sup>18</sup>F-DCFPyL will be included in the safety set.

#### **5.4.3.** Evaluable Set

*Evaluable subjects* in Cohort A are those who were dosed, had a prostatectomy or lymphadenectomy, and provided a <sup>18</sup>F-DCFPyL PET image result (positive or negative) and a corresponding histopathology result (positive or negative).

Evaluable subjects in Cohort B are those who were dosed, received a conventional image guided biopsy, and provided a <sup>18</sup>F-DCFPyL PET image result (positive or negative) and a corresponding histopathology result (positive for prostate cancer or negative), along with a conventional image that confirms the location of the histopathology sample.

#### 5.4.4. Change in Planned Protocol Procedure Set

The change in planned protocol procedure set includes dosed subjects in Cohort A who did not have a prostatectomy and lymphadenectomy due to change of planned management, and subjects in Cohort B who did not have conventional guided biopsy due to change of planned management. See figure 1 above for definition of change in planned management.

#### 5.4.5. Per Protocol Set

The Per-protocol set is defined as subjects in the Evaluable set without any major protocol deviations. Major protocol deviations will be identified prior to database lock and analysis.

#### 5.4.6. PK Blood Set

Subjects who provide at least six of the nine scheduled blood samples.

#### 5.4.7. PK Urine Set

Subjects who provided at least two of the three scheduled urine samples.

#### 5.5. Derived and Transformed Data

#### **5.5.1.** Baseline Definition

Baseline will be the latest pre-dose value.

#### 5.5.2. Baseline Age

Age is computed in the database as the number of full year increments from date of birth to informed consent date.

#### **5.5.3. Study Day**

Study day will be computed as the date of assessment minus the Dosing date (plus one if the assessment date is on or after the dose date).

#### 5.5.4. Change and Percent Change from Baseline

Change from baseline will be computed as any post baseline follow-up value minus the baseline value.

Percent change from baseline will be computed as 100 times the (post-baseline value minus the baseline value) divided by the baseline value. If the baseline value or the post-baseline value is missing, change from baseline and percent change from baseline will be missing.

#### **5.5.5.** Prior and Concomitant Medications

Prior medications are those administered prior to <sup>18</sup>F-DCFPyL administration date; concomitant medications are those administered from <sup>18</sup>F-DCFPyL administration through last study visit. If the concomitant medication does not have a full date then the algorithm in Section 5.6.2 will be used to determine if it is a pre- or post-dose medication.

#### **5.5.6.** Treatment-Emergent Adverse Events

Treatment emergent AEs are defined for all subjects as AEs occurring from the day of, but after <sup>18</sup>F-DCFPyL administration through the date prior to prostatectomy, lymphadenectomy, or change in planned procedure for subjects who underwent a procedure. For subjects who did not receive a procedure, TEAEs are collected up to 10 days after drug administration. For subjects in Cohort B who had a conventional imaging guided biopsy only, treatment emergent is defined as AEs occurring from the day of <sup>18</sup>F-DCFPyL administration through 28 days post biopsy.

### 5.5.7. Sensitivity, Specificity, PPV, and NPV

Sensitivity, specificity, PPV and NPV will be defined based on a <sup>18</sup>F-DCFPyL image result (positive or negative) and a histopathology result (positive or negative).

Table 3: Classification of <sup>18</sup>F-DCFPyL Imaging Result and Histopathology Result

| | Histopatho | | |
|-------------------------------------------------|-------------|------|------|
| <sup>18</sup> F-DCFPyL Image Positive* Negative | | | |
| Positive | TP | FP | I(p) |
| Negative | Negative FN | | I(n) |
| | R(p) | R(n) | N |

TP=true positive; FP=false positive; FN=false negative; TN=true negative.

The following statistics will be computed:

- Sensitivity = TP/R(p),
- Specificity = TN/R(n),
- Positive predictive value (PPV) = TP/I(p),
- Negative predictive value (NPV) = TN/I(n).

R(p) and R(n) denote the number of subjects with positive and negative histopathology results, respectively.

I(p) and I(n) denote the number of subjects with positive and negative <sup>18</sup>F-DCFPyL images, respectively.

N indicates the number of subjects

<sup>\*</sup>positive histology should be for prostate cancer only

### 5.5.7.1. Primary Endpoints and Pelvic Lymph Nodes

The primary endpoints of sensitivity and specificity are defined from lymph node imaging results and corresponding pelvic lymph node histology. For an imaging result to be deemed positive for this endpoint, the tissue must have first been removed from that corresponding area. This ensures that an imaging result has the ability to align with the results achieved from pathology. This will be applied to Cohort A subjects only.

PPV and NPV will also be calculated as secondary endpoints from the pelvic lymph nodes. The same definitions used below will apply.

| Criteria for Positive PyL Imaging Result | Criteria for Lymph Node Dissection and Positive Histology |
|---|---|
| If Right or Left Pelvic Lymph Nodes Minimum Template = Positive and • Tissue was removed from left template and total left nodes removed ≥1 and Template Left Pelvic LN Lesion Count | ≥1 positive lymph node on right template if Template Right Pelvic LN Lesion Count from imaging is ≥0 or ≥1 positive lymph nodes on left template if Template Left Pelvic LN Lesion Count from |
| ≥1 or • Tissue was removed from right template and total right nodes removed ≥1 and Template Right Pelvic LN Lesion Count ≥1 or Tissue was removed from Pre-sacral nodes and total pre-sacral nodes removed ≥1 and Pre-Sacral Pelvic LN Lesion Count ≥ 1 | imaging is ≥0 or ≥1 positive lymph nodes on pre-sacral nodes if Pre-Sacral Pelvic LN Lesion Count from imaging is ≥0 or ≥1positive lymph nodes on other pelvic lymph nodes if Other Pelvic Lymph Node Count from imaging is ≥0 |
| or Tissue was removed from Other lymph nodes and Total nodes removed >=1 and Other Pelvic LN Lesion Count ≥ 1 or | |

If tissue was removed from right template and total right nodes removed ≥1 and resection included tissue along the external iliac artery and Right pelvic lymph node external iliac artery= positive or

If tissue was removed from left template and total left nodes removed ≥1 and resection included tissue along the external iliac artery and left pelvic lymph node external iliac artery= positive or

If tissue was removed from right template and total right nodes removed ≥1 and resection included tissue along the common iliac vein and Right pelvic lymph node common iliac vein= positive or

If tissue was removed from left template and total left nodes removed ≥1 and resection included tissue along the common iliac vein and left pelvic lymph node common iliac vein=positive or

If tissue was removed from right template and total right nodes removed ≥1 and resection included tissue along the common iliac artery and Right pelvic lymph node common iliac artery= positive or

If tissue was removed from left template and total left nodes removed ≥1 and resection included tissue along the common iliac artery and left pelvic lymph node common iliac artery= positive

If Template Right Pelvic LN Lesion Count from imaging is  $\geq 0$  and Total number of positive lymph nodes from Right Template  $\geq 1$  or

If Template Left Pelvic LN Lesion Count from imaging is  $\geq 0$  and Total number of positive lymph nodes from Left Template  $\geq 1$ 

If any of the above criteria are met for imaging then PyL Imaging Result=Positive. If Cohort =A and lymphadenectomy was performed, and lesion counts from imaging results are available for at least one location (right, left, pre-sacral or other) but the above criteria are not met for imaging, then PyL Imaging Results = Negative.

If the above criteria for histology are met then Histology is positive. If all available positive lymph nodes=0 where the corresponding lesion count from imaging≥0 then Histology is negative.

If the lesion counts from all 4 locations (right, left, pre-sacral, and other lymph nodes) are not evaluable on imaging or tissue is not removed from all 4 locations then this endpoint will be missing.

#### **5.5.7.2.** Biopsy

Sensitivity and PPV are defined from imaging results in subjects undergoing a biopsy confirmed by conventional imaging and histology obtained from this biopsy. This will be performed for Cohort B only.

| Criteria for Positive PyL Imaging Result | Criteria for Biopsy and Positive Histology |
|---|---|
| Biopsied Lesion consistent with PSMA Positive uptake on the <sup>18</sup> F-DCFPyL PET/CT = yes | Pathology result=Positive for prostate cancer |

If Cohort =B, imaging and histology are obtained for the biopsy, and the above criteria are not met (Biopsied Lesion consistent with PSMA Positive uptake on the <sup>18</sup>F-DCFPyL PET/CT = no or pathology result = negative) then results = Negative for each respective endpoint.

#### 5.5.7.3. Prostate Gland

Sensitivity, specificity, PPV and NPV will be calculated from imaging and histology results from the prostate gland. This will be performed for subjects in Cohort A only.

| Criteria for Positive PyL Imaging Result | Criteria for Positive Histology |
|---|---|
| For category = PYL and Prostate gland right lesion count $\geq 1$ or Prostate gland left lesion count $\geq 1$ | If Prostate gland right lesion count ≥0 from imaging and Adenocarcinoma is present at right side of prostate or |
| | Prostate gland left lesion count ≥0 from imaging and Adenocarcinoma is present at left side of prostate |

If Cohort = A and Adenocarcinoma results are not missing for the right or left side of the prostate and the above criteria is not met, then result = Negative.

If imaging results are both not evaluable or the presence of adenocarcinoma is missing from both the left and right side of the prostate then this endpoint is missing.

#### 5.5.7.4. PPV for Changes in Planned Treatment

PPV will be calculated from imaging and histology results for the subset of subjects who had a change in the planned protocol procedure. Only a subset of these subjects may have tissue available for PPV.

| Criteria for Positive PyL Imaging Result | Criteria for Procedure and Positive<br>Histology |
|---|---|
|---|---|

| If subject in Cohort A and category=PYL and Is the 18F-DCFPyL PET/CT scan consistent with PSMA Positive cancer uptake = yes and Location of lesion count from imaging = location of lesion from histology and Lesion count for location >=1 from imaging | If Cohort A and prostatectomy and lymphadenectomy performed=no and Reason= Other, unscheduled Biopsy='Yes' and Pathology result=Positive for prostate cancer |
|---|---|
| If Cohort B and category = PYL and Prostate gland right lesion count $\geq 1$ or Prostate gland left lesion count $\geq 1$ | If Cohort B and Biopsy performed =no and Adenocarcinoma present at right or left side of prostate = yes |
| If Cohort B and category = PYL and positive imaging criteria from Section 5.5.7.1 is met. | If cohort B and biopsy performed = no and ≥1 positive lymph node on right or left template, pre-sacral nodes, or other pelvic lymph nodes |

The denominator of the above subset is the subset of subjects who had a change in the planned protocol procedure defined in Figure 1 and who had both imaging and histology results.

If imaging results are not evaluable then this endpoint is missing.

#### 5.5.8. Lesions Per Subject

The number of lesions detected on imaging categorized as bone, lymph nodes, soft tissue, and the prostate gland will be determined by each of the central imaging core lab independent readers. The sum of lesions per subject per tissue type and overall will be computed for each subject based on each reader's lesion count. This will be calculated from the <sup>18</sup>F-DCFPyL PET/CT scan results as well as the conventional imaging results.

| Bone | Soft Tissue | Lymph nodes | Prostate Gland |
|---|---|---|---|
| BN Skull | ST Brain | LN Cervical | ST Prostate Gland Left |
| BN Thorax | ST Neck | LN Supraclavicular | ST Prostate Gland Right |
| BN Spine | ST Lungs | LN Axillary | |
| BN Pelvis | ST Esophageal | LN Mediastinal | |
| BN Extremities | ST Liver | LN Hilar | |
| | ST Gall Bladder | LN Mesenteric | |
| | ST Spleen | LN Elbow | |
| | ST Pancreas | LN Popliteal | |
| | ST Adrenal | LN Peri-aortic/para-aortic | |
| | ST Kidney | LN Other, Non-Pelvic | |
| | ST Bladder | PLN Template Right | |
| | ST Prostate Bed | PLN Template Left | |
| | ST Seminal Vesicle | PLN Pre-Sacral | |
| | ST Skin | PLN Other, Pelvic | |
| | ST Muscle | | |
| | ST Other | | |

#### 5.5.9. Visit Windows

Data will be analyzed according to the nominal time points. Visit windows will not be used.

#### 5.5.10. Decay Corrected Dose at Time of Administration

The calculations in this section will need to be performed for the pre- and post- injection values for <sup>18</sup>F-DCFPyL administration as well as pre- and post- injection from the Syringe to the flask for reference values.

If a decay correction was performed for the pre-or post- dose values then Correction Factor =1. Otherwise:

```
 \text{Correction Factor} = e^{(\ln(2)*(pre\ or\ post\ injection\ time(min)-injection\ time\ (min)))}/_{110\ min}
```

where the above formula will be calculated for each of the following pre and post injection times:

pre-dose

post dose

syringe prior to flask syringe post flask

start of measurement times with each PK period

Convert all pre- and post- injection amounts to mCi: 37MBq = 1mCi

If there was no post decay correction then:

```
Decay Corrected Dose at time of Administration = (pre injection amount (mCi)*Correction Factor Pre Dose)- \frac{Post\ injection\ amount\ (mCi)}{Correction\ Factor\ Post\ Dose}
```

If there was a post decay correction then:

Decay Corrected Dose at time of Administration(mCi) = (pre injection amount(mCi) – post injection amount(mCi))

Calculate decay corrected doses at time of administration in both mCi for all subjects and MBq for all subjects.

The Decay corrected pre-injection Reference Standard of syringe prior to injection into flask = amount (μCi) in syringe prior to injection into flask\*Correction Factor of syringe prior to flask.

The Decay corrected post-injection Reference Standard of syringe after injection into flask = amount ( $\mu$ Ci) in syringe after injection into flask\*Correction Factor of syringe after flask.

The decay corrected reference standards are only needed in µCi.

#### 5.5.11. Lesion location defined from SUV values

There are three SUV values collected:  $SUV_{max}$ ,  $SUV_{peak}$  and  $SUV_{mean}$ . There are four locations that each of these SUV values could be present in: Bone, Soft tissue, prostate, and lymph nodes ('prostate gland right' and 'prostate gland left' were defined as a separate location from soft

tissue) as defined in Section 5.5.8. There are three reference values per subject at the following locations: Aorta, Liver and Muscle. For each tumor location that is not a reference location,  $SUV_R$  will be calculated against each reference as follows:

$$SUV_R = \frac{SUV_{MAX\_Tumor}}{SUV_{MEAN\_Re\ ference}}$$

Some subjects may have multiple SUV values within each location. These results will be averaged to derive one result per location and since there results should be similar per reviewer, only results for reviewer 1 will be used in any analyses. Subjects in Cohort B may have both a biopsied lesion and a tissue lesion within the same location. These SUV values should be summarized separately.

#### 5.5.12. Change in Clinical Management Plan from Questionnaire

A change in the Clinical Management plan from the pre-PyL scan assessment to the post-PyL scan assessment will be defined from any of the following questions:

- If there is a change in planned diagnostic biopsy from pre-PyL to post-PyL
- If there is a change in planned surgery from pre-PyL to post-PyL
- If type of surgery planned pre-PyL does not match post-PyL
- If type of planned chemotherapy changes from pre-PyL to post-PyL
- If there is a change in planned other immunotherapy/investigational therapy from pre-PyL to post-PyL
- If planned radiation therapy changed from pre-PyL to post-PyL
- If chemotherapy plan changed from pre-PyL to post-PyL
- If hormonal/ADT plan changed from pre-PyL to post-PyL
- If there is a change in other therapy/intervention from pre-PyL to post-PyL

An overall change score will be calculated as well as a change in each of the above criteria alone.

#### **5.5.13. PSA groups**

PSA will be categorized into the following groups:

| <0.2 ng/mL |
|-------------------|
| 0.2 to <4.0 ng/mL |
| 4 to <20.0 ng/mL |
| 20.0 to <50.0 |
| ng/mL |
| ≥50 ng/mL |

#### 5.5.14. Gleason Scores

The Gleason score will be derived by concatenating the primary Gleason grade to the secondary Gleason grade, separated by a plus sign (e.g., 3+4). The total Gleason score will be computed as the sum of the primary and secondary Gleason grades (7 in the example of 3+4 provided here).

Gleason Score from prostatectomy will be categorized into the following groups as shown in the table based on the sum of primary and secondary Gleason Grades:

| Primary Gleason Grade | Secondary Gleason Grade | Total |
|-----------------------|-------------------------|-------|
| 3 | 3 | ≤ 6 |
| 3 | 4 | 7 |
| 4 | 3 | 7 |
| 4 | 4 | 8 |
| 4 | 5 | 9 |
| 5 | 5 | 10 |

#### **5.5.15.** Prior Prostate Cancer History and Therapies

If any of the follow variables have partial dates where only month and year are present, then months will be calculated as ((dose year - parameter year) x12) + ((dose month-parameter month) +1). Otherwise, with full dates, the calculation would be as follows:

Months since last prostate cancer staging = (Dose date – prior prostate cancer staging date)/30.4.

Months from Prior Therapy to Dose =  $(Dose\ Date - Prior\ prostate\ Therapy\ stop\ date)/30.4$ 

Months from Prior Radiation to Dose= (*Dose Date – Prior radiation Therapy stop date*)/30.4

Months from Prior Surgery to Dose =  $(Dose\ Date - Prior\ prostate\ surgery\ date)/30.4$ 

Months from Staging to Dose= (Dose Date – Primary tumor staging date)/30.4

Months since last Prior Therapy to Dose = (Dose Date – Prior therapy date)/30.4.

Full dates must be present for duration variables below:

Duration of Prior Therapy (days) = (Prior Prostate Therapy stop date – Prior prostate therapy start date) +1.

Duration of Prior Radiation Therapy (days) = (Prior Radiation Therapy stop date - Prior Radiation therapy start date) +1

#### 5.5.16. Estimate GFR

Estimate GFR (eGFR) will be calculated using the Modification of Diet in Renal Disease (MDRD) Equation<sup>4</sup>:

eGFR (mL/min/1.73 m<sup>2</sup>) =  $175 \times (S_{cr})^{-1.154} \times (Age in years)^{-0.203} \times (0.742 if female) \times (1.212 if African American)$ 

Where Scr= Serum creatinine (mg/dL)

#### 5.5.17. Renal impairment

If Estimated GFR  $\geq$ 90 then Normal (no impairment), otherwise if  $0 \leq$ eGFR $\leq$ 90 then Abnormal.

## **5.5.18.** Laboratory Parameter Unit Conversions

| Lab Parameter | Original<br>Unit | Conversion<br>Factor (multiply) | Final SI<br>Unit |
|---|---|---|---|
| ALT, Alkaline Phosphatase | U/L | 0.0167 | Ukat/L |
| Albumin, Total Protein, hemoglobin | g/dL | 10 | g/L |
| BUN | mg/dL | 0.357 | mmol/L |
| Calcium | mg/dL | 0.25 | mmol/L |
| Chloride, Potassium, Sodium | mEq/L | 1 | mmol/L |
| Creatinine | mg/dL | 88.4 | umol/L |
| Glucose | mg/dL | 0.0555 | mmol/L |
| Total Bilirubin | mg/dL | 17.104 | umol/L |
| Total Testosterone | ng/dL | 0.0347 | nmol/L |
| Total Testosterone | ng/mL | 3.4672 | nmol/L |
| Triglycerides | mg/dL | 0.0113 | mmol/L |
| Hematocrit | % | 0.01 | L/L |
| Basophils, Eosinophils, lymphocytes, monocytes, neutrophils, platelets, WBC count | k/cumm | 1 | 10 <sup>9</sup> /L |
| Basophils, Eosinophils, lymphocytes, monocytes, neutrophils, platelets, WBC count | k/μL | 1 | 10 <sup>9</sup> /L |
| Basophils, Eosinophils, lymphocytes, monocytes, neutrophils, platelets, WBC count | $10^3/\mu$ L | 1 | 10 <sup>9</sup> /L |
| Basophils, Eosinophils, lymphocytes, monocytes, neutrophils, platelets, WBC count | 10 <sup>9</sup> /L | 1 | 10 <sup>9</sup> /L |

| Basophils, Eosinophils, lymphocytes, monocytes, neutrophils, platelets, WBC count | k/mcl | 1 | 10 <sup>9</sup> /L |
|---|---|---|---|
| RBC Count | m/mcl | 1 | $10^{12}/L$ |
| RBC Count | m/µL | 1 | $10^{12}/L$ |
| RBC Count | mil/cumm | 1 | $10^{12}/L$ |
| RBC Count | 10 <sup>12</sup> /L | 1 | $10^{12}/L$ |
| RBC Count | $10^{12}/L$ | 1 | $10^{12}/L$ |
| RBC Count | $10^6/\mu L$ | 1 | $10^{12}/L$ |
| PSA | ng/mL | 1 | ug/L |

## 5.6. Handling of Missing Data

### **5.6.1.** Missing Efficacy Endpoints

No imputation methods will be employed.

## 5.6.2. Missing Start and Stop Dates for Concomitant Medication

Partial or missing medication start, and end dates will be categorized as occurring prior to or after dose using the following logic. If a medication categorized as post-dose had a start date< dose date or a start year <dose year or a start year=dose year and start month<dose month then it will be summarized as both a pre- and post- medication.

| Start Date | Stop Date | Category |
|---|---|---|
| < dose date or Year< dose year or year= dose year and | date< dose date or year <dose and<="" or="" td="" year=""><td>Pre-dose</td></dose> | Pre-dose |
| month< dose month or | month <dose month<="" td=""><td></td></dose> | |
| year=dose year or date=missing | | |
| < dose date or Year< dose year or year= dose year and | Missing or date< dose date or year <dose or="" year="dose&lt;/td"><td>Pre-Dose</td></dose> | Pre-Dose |
| month< dose month | year and month <dose month="" or="" td="" year="dose" year<=""><td></td></dose> | |
| Year = dose year and month<br>= dose month and day is<br>missing | Year = dose year and month < dose month | Pre-dose |
| >dose date or year=dose year and month dose month | missing | Post Dose |
| >dose date or year=dose year and month> dose month | | Post Dose |
| | ≥ dose date or year>dose year<br>or year=dose year and month ≥<br>dose month | Post Dose |
| Date <dose and="" date="" dose="" month<="" month≤dose="" or="" td="" year="" ≤=""><td>Year=dose year and month=dose month</td><td>Post Dose</td></dose> | Year=dose year and month=dose month | Post Dose |
| Missing | missing | Post Dose |
| < dose date or Year< dose | ≥ dose date or year>dose year | Pre and Post Dose |
| year or year= dose year and | or year=dose year and month ≥ | |
| month< dose month | dose month | |

#### 6. STUDY POPULATION

## 6.1. Disposition

Subject disposition will display the number of consented subjects and the percentage of them who failed screening. The number of subjects in the safety analysis set as well as the number and percentage of subjects in the evaluable set, per-protocol set, change in planned protocol procedure set, and PK sets will also be summarized. The number and percentage of subjects who completed or discontinued from the study with the reason for discontinuation, will be tabulated. All percentages for discontinuation reasons will be based on the number of subjects in the safety population.

#### **6.2.** Protocol Deviations

Protocol deviations will be summarized in the clinical study report based on the protocol deviation log.

Protocol deviations will be listed, including their classification as major or minor for the Safety Set.

## 6.3. Demographic and Baseline Characteristics

Demographic and baseline characteristics: age at informed consent in years, categorical age (<65 years, ≥65 years), race, ethnicity, height in cm, weight in kg, and BMI in kg/m² will be summarized by cohort for the safety set, the evaluable set, and the per protocol set.

## 6.4. Medical History, including Prostate Cancer History

Medical history will be summarized by MedDRA system organ class (SOC) and preferred term (PT) using frequencies and percentages.

Prior prostate cancer history will also be summarized using summary statistics for months since most recent prostate cancer staging, PSA (ng/mL) and testosterone (ng/dL). Frequencies and percentages will be presented for whether PSA results were captured within 30 days from Baseline, PSA groups, primary Gleason grade, secondary Gleason grade, Gleason total score, primary tumor stage (T), regional lymph node stage (N), distant metastasis stage (M) and renal impairment status.

Medical history and prostate cancer history will be presented for the safety set, the evaluable set and the per-protocol set.

## **6.5.** Prior Prostate Cancer Therapies and Surgeries

For prior prostate cancer therapies, each line of therapy is captured into a group ranging from A-O, where A is the first line of therapy and O is the last line of therapy. The drugs within each are collected. Prior to locking the database, these drugs will be categorized into groups. An additional categorization will also be performed to show types of prostate cancer therapies. These therapies will be summarized overall for the drugs within the different lines of therapies. The number of therapy regimens received, and types of prostate cancer therapies will be summarized.

Progenics Pharmaceuticals, Inc. Statistical Analysis Plan – Protocol PyL-2301

September 5, 2018

Radiation therapy will be presented to show whether it was prostate related or not, and radiated site.

Months since last reported surgery will also be summarized. Surgeries will also be presented by system organ class and preferred term.

All prior prostate cancer therapies and surgeries will be presented for the safety set, the evaluable set and the per protocol set.

## 6.6. Prior Medication History and Medications Present at Entry

Prior medications will be summarized by ATC4 class and generic name using frequencies and percentages. Prior medications will also be listed.

Prior medication history will be presented for the safety set, the evaluable set and the per protocol set.

## 6.7. Conventional Imaging at Baseline

Type of bone scans, bone scans obtained within 10 hours of dosing, MRI/CT performed, and type of MRI/CT will be summarized by the safety set, the evaluable set and the per protocol set.

#### 7. EFFICACY

#### 7.1. General Considerations

Statistical tests and their corresponding confidence intervals will be two-sided at the 0.05 significance level.

The estimation of sensitivity and specificity rely on the central imaging core lab independent readers. Each reader's assessments will be summarized separately.

## 7.2. Testing Statistical Assumptions Including Comparability at Baseline

#### 7.2.1. Test of Proportions

The assumption underlying the normal approximation to the binomial distribution, used in the computation of confidence intervals for sensitivity, specificity, PPV, and NPV, is that the sample size is such that np>5 and n(1-p)>5, where n is the sample size and p is the binomial probability. It is expected that the sample size for each statistic will be sufficient to meet this assumption. In the event that the sample size is not sufficient, Agresti-Coull exact tests will be used. As there is only one treatment in this study, there will be no testing of baseline comparability.

#### 7.2.2. Test of means

The assumption of normality of the data may be violated when testing for differences in means. If data fail the Shapiro-Wilk test for normality within each group, then a Wilcoxon rank sum test will be used for the comparison of 2 groups and a Kruskal-Wallis test for comparison of 3 groups to test for differences in the distribution between groups. For 2 group comparisons, an exact 95% confidence interval will be generated for the difference scores. For a 1-way repeated

measures ANOVA, if the assumption of normality is not met then a Friedman test will be performed.

### 7.3. Statement of the Null and Alternate Hypotheses

The null and alternative hypotheses are stated in Section 4.3.

## 7.4. Subgroup Analyses

No subgroup analyses are planned, but they may be examined for exploratory purposes.

## 7.5. Multiple Comparisons and Multiplicity

Within Cohort A, the type I error rate will be preserved by requiring that both null hypotheses be rejected in order to draw the conclusion that <sup>18</sup>F-DCFPyL is efficacious for imaging. In addition, the three readers from the central imaging core laboratory are independent and requiring that the same 2 of 3 readers agree about sensitivity and specificity (Cohort A) will control for type I error.

## 7.6. Analysis of the Primary Efficacy Endpoint

### 7.6.1. Primary Efficacy Analysis of Primary Endpoints

The primary analysis for subjects in Cohort A will be addressed by computing point estimates and 95% two-sided confidence intervals (CIs) for specificity first and if the null hypothesis is rejected for specificity then sensitivity will be tested next. Both outcomes are assessed on the subject level (one overall outcome per subject) in the *evaluable set*. If the *per protocol* set exists, then this analysis will be performed on the *per protocol* set as a supplemental analysis. The normal approximation to the binomial distribution is planned assuming the assumptions have been met (See Section 7.2). Sensitivity and specificity will be computed for each of three central imaging core lab independent PET/CT readers.

The null hypothesis for specificity will be rejected if the lower limit of the 95% CI exceeds 80% for at least two of the three independent central PET/CT readers. If statistical significance is achieved for specificity where the null hypothesis is rejected, then sensitivity will be tested where the null hypothesis will be rejected if the lower limit of the 95% CI exceeds 40% for the same two readers who rejected the null hypothesis for specificity.

#### 7.6.2. Sensitivity Analyses of the Primary Endpoints

A sensitivity analysis of the primary endpoint will be performed allowing any 2 of the 3 central PET/CT readers to reject the null hypothesis for sensitivity only after specificity has been deemed a success. This analysis will require agreement of at least 2 readers, but they do not need to be the same 2 central readers to reject the null hypothesis for specificity and sensitivity. This analysis will be performed for the evaluable and per protocol sets.

## 7.7. Analysis of Secondary Efficacy Endpoints

Analysis of secondary efficacy endpoints will be conducted regardless of the outcomes of the primary analyses. Diagnostic testing and imaging detection rates will be analyzed for the evaluable set. The PK parameters will be summarized for the PK blood set.

#### 7.7.1. NPV and PPV in Cohort A

Point estimates and two-sided 95% CIs for PPV and NPV will be computed for the prostate gland and the lymph nodes in Cohort A subjects in the Evaluable Set. The normal approximation to the binomial distribution is planned assuming the assumptions have been met (See Section 7.2). PPV and NPV will be computed for each of the three central imaging core lab independent PET/CT readers.

#### 7.7.2. PPV and Sensitivity in Cohort B

Point estimates and two-sided 95% CIs for PPV and Sensitivity will be computed from the conventional guided biopsy obtained from subjects in Cohort B for the Evaluable Set. The normal approximation to the binomial distribution is planned assuming a null hypothesis of 0.5. If the assumptions are not met, then confidence intervals derived from an Agresti-Coull exact test will be used (See Section 7.2). Results will be computed for each of the three central imaging core lab independent readers.

#### 7.7.3. Detection Rates for Lesion Counts in both Cohorts Combined

For subjects in Cohort A and B combined, the sum of the lesions per tissue type and overall per subject will be summarized showing the N, mean, median, standard deviation, minimum and maximum values for each central imaging core lab reader including the reader of conventional scans. <sup>18</sup>F-DCFPyL images and conventional images will be summarized separately and the mean of each reader's results from <sup>18</sup>F-DCFPyL PET/CT will be compared to conventional imaging using a one-way repeated measures ANOVA. If the assumptions are not met for this test (see Section 7.2), then a Friedman's test will be performed to determine if there is a difference between any of the groups. If significant is determined from either the ANOVA or the Friedman's test, then a Dunnett's test will be performed to show where the difference exists between each reviewer and the conventional scan. A p-value and 95% confidence interval for the difference in means will be presented for each <sup>18</sup>F-DCFPyL PET/CT reviewer versus conventional imaging. This analysis will be performed on the Evaluable Set.

#### 7.7.4. PK

Blood, plasma, and urine collection at each nominal time will be collected twice per patient. The mean of the values at each nominal time will be used in the creation of parameters used in the analysis. For each subject, blood concentration-time data using actual blood draw times rather than nominal times will be computed by non-compartmental analysis and pharmacokinetic parameters will be generated. Additional blood concentration-time data will be fitted into a two-compartment model to calculate  $T_{1/2\text{-alpha}}$  and  $T_{1/2\text{-beta}}$ . Summary statistics for blood will be presented for maximum concentration ( $C_{max}$ ), area under the (activity-time) curve (AUC), body weight normalized clearance (CL), volume of distribution at steady-state ( $V_{ss}$ ), time to maximum concentration ( $T_{max}$ ), half-life( $T_{1/2}$ ) [noncompartmental analysis],  $T_{1/2}$ -alpha and  $T_{1/2}$ -beta [2-

compartment modelling], and mean residence time (MRT). Since there are two values collected per nominal time, the mean of these values within nominal time will be derived prior to generating the PK parameters. These PK parameters will be derived by an external analyst then summarized for the PK blood set. PSA groups, eGFR groups and eGFR will also be summarized for the PK blood set.

Summary statistics for urinary excretion will be presented for Tmax, Rate max, Rate last, T1/2elim, and Cumulative Urine Recovery. For % of injected dose recovered per each urine collection interval per subject will be used to calculate Tmax, Rate max, Rate last, T<sub>1/2elim</sub>, and cumulative urine recovery by 4 and 8 hours post-administration if feasible. These PK parameters will be derived by an external analyst then summarized for the PK urine set. eGFR groups as defined in Section 5.5.16 and eGFR will also be summarized for the PK urine set.

The ratio of plasma-to-blood concentrations will be calculated per subject/time-point.

#### 7.8. Analysis of Exploratory Endpoints

Sensitivity and specificity of the prostate gland as well as  $SUV_{max}$ ,  $SUV_{peak}$  and  $SUV_r$  will all be analyzed on the evaluable set. Change in Management defined from the questionnaire will be summarized on the safety set. The PPV endpoint will be analyzed on the Change in Planned Protocol Procedure Set.

- SUV<sub>max</sub>, SUV<sub>peak</sub>, SUV<sub>mean</sub>, and volume will be summarized for each tissue location (bone, lymph nodes, soft tissue, and prostate gland) and each of the 3 central imaging core lab independent readers using the evaluable set from both cohorts. SUV<sub>r</sub> will be summarized in the same manner including a reference lesion also. A 95% confidence interval for the mean or distribution will be presented for each reader based on the assumption on normality defined in Section 7.2.
- Differences in the average across all 3 reviewers for SUV<sub>max</sub>, SUV<sub>peak</sub>, SUV<sub>r</sub>, SUV<sub>mean</sub>, and volume will be compared between histology outcomes using a t-test that assumes unequal variances. If the assumptions for the t-test are not met then a Wilcoxon rank sum test will be performed with corresponding exact 95% confidence intervals defined in section 7.2.
- The average SUV<sub>max</sub>, SUV<sub>peak</sub>, SUV<sub>r</sub>, SUV<sub>mean</sub>, and volume values across all reviewers will be compared between Gleason Score groups at time of radical prostatectomy, Baseline PSA groups and testosterone groups split at the median value. The comparisons of means between groups will be performed using a generalized linear model. If normality cannot be assumed then a Kruskal-Wallis test will be performed instead. Within each group a 95% confidence interval will be presented.
- Point estimates and two-sided 95% CIs for Specificity and Sensitivity will be computed from the prostate gland for Cohort A in the Evaluable Set. The normal approximation to the binomial distribution is planned assuming a null hypothesis of 0.5. If the assumptions are not met then confidence intervals derived from an Agresti-Coull exact test will be used (See Section 7.2). Results will be computed for each of the 3 central imaging core lab independent readers.

- Clinical management questions pre- and post <sup>18</sup>F-DCFPyL PET/CT imaging will be summarized from the questionnaire evaluated by a central reader. The proportion of subjects in Cohort A who had a change in intended clinical management plan from pre-to post PyL scans will be analyzed using a one sample binomial test.
- Point estimates and two-sided 95% CIs for PPV will be computed for the change of management set. An Agresti-Coull 95% confidence interval will be used will be used assuming a null hypothesis of 0.5. Results will be computed for each of the 3 central imaging core lab independent readers.

## 7.9. Reader Reliability

There are four imaging readers who were trained to perform our central reads used in much of the analyses. Only three of these readers will perform these reads with the fourth reader as an alternative if needed. Variability of these readers regarding the primary endpoint for the evaluable set will be tested as described below. The following is assumed:

N<sub>i</sub>=total number of subjects with the primary endpoint in the evaluable set (i=1, 2,...N)

K=number of readers (3)

 $R_i$ = number of responses (i=1,2)

n<sub>ij</sub>=number of times subject i is in response group j

#### 7.9.1. Intra-Reader Reliability

Prior to reading any images, a random subset of 30 PyL images will be randomly selected by the Imaging vendor. Once the reads start, this subset will be re-introduced to each reader no sooner than 3 weeks after the original read. They will be read under identical conditions as the original read (same criteria evaluation, same analysis reporting, same analysis platform). The rate of agreement between the original reads and the re-reads for the primary endpoint in this subset will be compared using the intra-rater variability defined from Cohen's Kappa<sup>5</sup>. This calculation will be performed for each reader separately.

Cohen's Kappa = 
$$\frac{p_{a-}p_e}{(1-p_e)}$$
where  $p_a = \sum_{j=1}^R \frac{n_{jj}}{n}$ 

$$p_e = \sum_{j=1}^R \frac{n_{j+}}{n} \frac{n_{+j}}{n}$$

The standard error of Kappa  $\sigma_k\,\underline{w}ill$  be calculated as:

$$\sigma_{k} = \sqrt{\frac{P_{a}(1-P_{a})}{N(1-P_{e})^{2}}}$$

It is assumed that the concordance rate between time points for each reader will be at minimum of 93% with a Kappa of 86%. This would yield a 95% confidence interval of (0.68, 1) for a sample of 30 subjects.

#### 7.9.2. Inter-Reader Reliability

For the primary analysis of the primary endpoint the inter-reader reliability will be estimated using the multiple-reader generalized kappa statistic developed by Fleiss<sup>6,7</sup>.

$$Kappa = \frac{\bar{p} - \bar{p}_e}{1 - \bar{p}_e}$$

Variance: 
$$\frac{2}{NK(K-1)} \frac{\sum_{j=1}^{R} p_j^2 + (\sum_{j=1}^{R} p_j^2)^2 - 2\sum_{j=1}^{R} p_j^3}{(1 - \sum_{j=1}^{R} p_j^2)^2}$$

Where

$$p_j = \frac{1}{NK} \sum_{i=1}^{N} n_{ij}$$

$$p_i = \frac{\sum_{j=1}^{R} n_{ij} (n_{ij} - 1)/2}{K(K-1)/2}$$

$$\bar{p} = \frac{\sum_{i=1}^{N} p_i}{N}$$
 (overall agreement)

$$\bar{p}_e = \sum_{j=1}^R p_j^2$$
 (expected chance agreement)

The generalized Kappa statistic and a 95% confidence interval will be computed.

#### 8. SAFETY AND TOLERABILITY

All safety data will be summarized by cohort.

# 8.1. Adverse Event Preferred Term and System Organ Class Summary Tables

An overall summary of frequency and percentage of treatment-emergent adverse events (TEAEs), most frequent (>5%) overall TEAEs, serious TEAEs, severe TEAEs (grade  $\geq$  3), TEAEs by grade, and treatment-related TEAEs will be presented by cohort and overall using the safety set.

#### 8.1.1. Summaries of Adverse Event Incidence Rates for All Subjects

Treatment-emergent adverse events will be summarized by SOC and PT using the frequency and percentage of subjects experiencing any adverse event, experiencing each SOC and experiencing each PT within each SOC, using the safety set. The number of occurrences of each adverse event will be included.

Treatment-emergent adverse events will be summarized by severity and for subjects who report adverse events with severity grades 3 or higher. The most severe occurrence of each event will be summarized by SOC and PT using the frequency and percentage of subjects experiencing any adverse event, experiencing each SOC and experiencing each PT within each SOC by cohort and overall, using the safety analysis set.

Treatment-emergent adverse events will be summarized by relationship to study drug. The most closely related occurrence of each event will be summarized by SOC and PT using the frequency and percentage of subjects experiencing any adverse event, experiencing each SOC and experiencing each PT within each SOC by cohort and overall, using the safety analysis set.

# 8.1.2. Summaries of Adverse Incidence Rates for Serious Adverse Events (SAE), Adverse Event Discontinuations, and Death

The overall summary table includes incidences of serious adverse events, adverse events that led to discontinuation and deaths.

Separate listings for serious adverse events, adverse events that led to discontinuation and deaths will be created.

## 8.2. Exposure to Study Drug

Exposure to study drug will be summarized using summary statistics for volume administered, location of injection, correction factor at pre and post dose, the decay corrected dose in mCi and MBq at time of administration, and any dose change due to an AE for the safety set.

#### **8.3.** Concomitant and Other Medications

Concomitant medications will be summarized by ATC4 class and generic term using frequencies and percentages for the safety analysis set.

### **8.4.** Routine Laboratory Data

Summary statistics for observed and change from baseline values of each laboratory analyte will be presented by visit for the safety set. Labs will include hematology and chemistry. A shift table will also be presented showing the shift in values from Baseline to follow up (below LLN, within LLN and ULN, above ULN, and missing). The following parameters will be created and summarized also:

Leukocytes = sum of Basophils, Eosinophils, Lymphocytes, Monocytes, and Neutrophils

Basophils/leukocytes = (Basophils/leukocytes)\*100

Eosinophils/leukocytes = (Eosinophils /leukocytes)\*100

Lymphocytes/leukocytes = (Lymphocytes /leukocytes)\*100

Monocytes/leukocytes = (Monocytes /leukocytes)\*100

Neutrophils/leukocytes = (Neutrophils /leukocytes)\*100

## 8.5. Vital Signs

Summary statistics for observed and change from baseline values of each vital sign (systolic and diastolic blood pressures, heart rate, respiratory rate, and temperature) will be presented by visit and cohort for the safety set.

#### **8.6.** ECG

Summary statistics for observed and change from baseline values of each ECG parameter will be presented by visit and cohort using the safety set. For QT interval, adjudicated QTc-Bazett and adjudicated QTc-Fidericia, the following groups will be summarized at Baseline and the pre-imaging visit: values above 450, above 480 and above 500. For these same parameters the following will be summarized at the pre-imaging time point only: Increase 31-50, increase >60, decrease 31-60, and decrease >60.

#### 8.7. Physical Examination

Not applicable

#### 9. PHARMACOKINETICS

Summary statistics for blood will be presented for maximum concentration (Cmax), area under the (activity-time) curve (AUC), clearance (CL), volume of distribution at steady-state (Vss), time to maximum concentration (Tmax), half-life(T1/2) [noncompartmental analysis], T1/2-alpha and T1/2-beta [2-compartment modelling], and mean residence time (MRT). Clearance and Vss will be body-weight normalized.

Percent of dose recovered in urine will be presented by collection intervals for the PK urine set. The following urinary kinetics will also be presented for this set: Tmax, Rate max, Rate last,  $T_{1/2}$  elim, and cumulative urine recovery by 4 and 8 hours post administration as % injected dose. The ratio of plasma-to-blood concentrations will be calculated per each subject/time-point.

#### 9.1. Derived Data

- Concentration of Reference Standard, µCi/mL =
  - (Decay Corrected pre injection reference standard of syringe prior to injection into flask—Decay Corrected post injection reference standard of syringe after injection into flask)/1000mL.
- Reference Standard CPM = <sup>18</sup>F-DCFPyL reference standard (CPM) from PK\*Decay Correction factor for measurement time defined for 0-4 hours
- Average CPM for Reference standard= Average of 3 CPM results collected for <sup>18</sup>F-DCFPyL std for 0-4 hours.
- Average CPM/ml for reference standard= Average CPM for reference standard/0.3
- Concentration of Reference Standard in CPM/ $\mu$ Ci = Average CPM/ml for reference standard/concentration of reference standard ( $\mu$ Ci/mL)
- For each blood, plasma and urine sample time, calculate:
  - $^{18}$ F-DCFPyL CPM<sub>b</sub> =  $^{18}$ F-DCFPyL CPM result at sample time\*correction factor for measurement time defined for the PK period the sample is drawn in
  - $CPM_b(ml) = CPM_b/0.3$

- CPM concentration( $\mu$ Ci/ml) = CPM<sub>b</sub> (ml) / Concentration of Sample in CPM ( $\mu$ Ci)
- Average CPM  $\mu$ Ci/ml = average CPM  $\mu$ Ci/ml within each unique nominal time
- Ratio of plasma to blood = Average CPM ( $\mu$ Ci/ml) for plasma/ Average CPM ( $\mu$ Ci/ml) for blood per unique sample nominal time
- For each urine sample, calculate:
  - Radioactivity excreted per collection interval ( $\mu$ Ci) = CPM ( $\mu$ Ci/ml) from urine\*urine collection volume (ml)
  - % Dose excreted = (Sum of Radioactivity exerted per collection interval( $\mu$ Ci) /(administered dose(mCi)\*1000))\*100
  - Average % dose excreted = average of individual % dose excreted per unique urine collection interval
  - Cumulative Average % dose excreted = sum of average % dose excreted over all unique urine collection intervals:
    - 0-4 hours = sum of average % dose excreted over 0-2 and 2-4 hours urine collection intervals
    - 0-8 hours = sum of average % dose excreted over all unique 0-2 and 2-4 hours urine collection intervals (0-2, 2-4, and 4-8 hours)

\_

Pharmacokinetic analyses will be conducted on pooled cohorts using the PK blood set and PK urine set.

# 10. PLANNED TREATMENT SAP CHANGES THAT DIFFER FROM THE PROTOCOL

- Screened population renamed to consented population as the definition states all subjects need to provide consent and not screening data.
- The Evaluable set was updated to state that subjects in Cohort A are required to have a prostatectomy and lymphadenectomy.
- The Change in Planned Protocol Procedure Set was added as a subject population to capture the subjects who had a change in the planned protocol procedure.
- The PK Evaluable set was divided into two groups: The PK Blood Set and the PK Urine set, as a subject could meet the criteria for one of these, but not the other.
- 'PPV of 18F-DCFPyL PET/CT imaging in subjects with corresponding histopathology that is outside the planned protocol surgical template or biopsy site' was updated to 'PPV of 18F-DCFPyL PET/CT imaging in subjects with corresponding histopathology for subjects who had a change in planned treatment per Cohort assignment'. Subjects may undergo a planned protocol procedure defined per the other cohort.
- The number of lesions per subject plotted against PSA and baseline testosterone for each of the 3 central imaging core lab readers will no longer be performed.
- SUV<sub>max</sub>, SUV<sub>peak</sub>, SUV<sub>r</sub> will no longer be summarized by subgroups: Previous radiation therapy (yes/no), Previous hormonal therapy (yes/no), or Previous chemotherapy (yes/no). Most subjects will be from cohort B only.
- Sensitivity will no longer be summarized by previous radiation therapy, previous hormonal therapy or previous chemotherapy. Since it is no longer the primary endpoint and it's not appropriate to combine cohorts for this analysis, it is no longer of interest.
- The following was added for PK: Additional blood concentration time data will be fitted into a two-compartmental model to calculate T<sub>1/2-alpha</sub> and T<sub>1/2-beta</sub>. For % of injected dose recovered per each urine collection interval per subject will be used to calculate Tmax, Rate max, Rate last, T<sub>1/2elim</sub>, and cumulative urine recovery if feasible.

#### 11. REFERENCES

- 1. ICH E6: Good Clinical Practice: Consolidated Guidance
- 2. ICH E9: Statistical Principles for Clinical Trials
- 3. Fleiss, J. L.; Levin, B.; Paik, M.C. (2003). Statistical Methods for Rates and Proportions (3rd ed.). New York: John Wiley & Sons
- 4. Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF, 3rd, Feldman HI, et al. A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009;150(9):604-12
- 5. Gwet, K.; Intrarater Reliability. Wiley Encyclopedia of Clinical Trials, Copyright 2008 John Wiley & Sons, Inc.

- 6. Woolson, R.; Statistical Methods for the Analysis of Biomedical Data. Copywright 1987 John Wiley & Sons, Inc.
- 7. Fleiss, J. L., Nee, J. C. M., and Landis, J. R. Ž1979. The large sample variance of kappa in the case of different sets of raters. *Psychol. Bull.*, 86, 974\_977.

## 12. APPENDIX

## 12.1. Table of Contents for Data Display Specifications

Table 4 contains a list of tables, listings and figures proposed for this study.

**Table 4: List of Tables, Listings and Figures** 

| Number | Title |
|---|---|
| 14.1-1 | Subject Enrollment and Disposition, Consented Subjects |
| 14.1.1: Baseline Summaries – Safety Set | |
| 14.1.1-1 | Demographics and Baseline Characteristics, Safety Set |
| 14.1.1-2 | Prostate Cancer History, Safety Set |
| 14.1.1-3 | Medical History, Safety Set |
| 14.1.1-4 | Prior Prostate Cancer Therapies, Safety Set |
| 14.1.1-5 | Prior Surgery, Safety Set |
| 14.1.1-6 | Conventional Imaging at Baseline, Safety Set |
| 14.1.1-7 | Baseline Medication Use, Safety Set |
| 14.1.2: Ba | seline Summaries – Evaluable Set |
| 14.1.2-1 | Demographics and Baseline Characteristics, Evaluable Set |
| 14.1.2-2 | Prostate Cancer History, Evaluable Set |
| 14.1.2-3 | Medical History, Evaluable Set |
| 14.1.2-4 | Prior Prostate Cancer Therapies, Evaluable Set |
| 14.1.2-5 | Prior Surgery, Evaluable Set |
| 14.1.2-6 | Conventional Imaging at Baseline, Evaluable Set |
| 14.1.2-7 | Baseline Medication Use, Evaluable Set |
| 14.1.3: Ba | seline Summaries – Per Protocol Set |
| 14.1.3-1 | Demographics and Baseline Characteristics, Per Protocol Set |
| 14.1.3-2 | Prostate Cancer History, Per Protocol Set |
| 14.1.3-3 | Medical History, Per Protocol Set |
| 14.1.3-4 | Prior Prostate Cancer Therapies, Per Protocol Set |
| 14.1.3-5 | Prior Surgery, Per Protocol Set |
| 14.1.3-6 | Conventional Imaging at Baseline, Per Protocol Set |
| 14.1.3-7 | Baseline Medication Use, Per Protocol Set |
| 14.2.1: Pr | imary Efficacy – Evaluable Set |
| 14.2.1-1 | Sensitivity and Specificity of the Pelvic Lymph Nodes for the Subjects in Cohort A, Evaluable Set |

| 14.2.2: Secondary Efficacy- Evaluable Set or PK Serum Set | |
|---|---|
| 14.2.2-1 | Diagnostic Testing for Secondary Endpoints, Evaluable Set |
| 14.2.2-2 | Summary of Imaging Detection Rates for Lesion Counts by Region- Evaluable Set |
| 14.2.2-3 | Summary of Pharmacokinetic Parameters for Cycle 1, Day1- PK Blood Set |
| 14.2.3: Ex | ploratory Efficacy |
| 14.2.3-1 | SUV Responses at Baseline- Evaluable Set |
| 14.2.3-2 | SUVR Responses at Baseline – Evaluable Set |
| 14.2.3-3 | SUV Responses by Histology Outcomes- Evaluable Set |
| 14.2.3-4 | SUV Responses and Volume at Baseline by PSA Groups- Evaluable Set |
| 14.2.3-5 | SUV Responses and Volume at Baseline by Gleason Score Groups at Time of Prostatectomy- Evaluable Set |
| 14.2.3-6 | SUV Responses and Volume at Baseline by Testosterone Groups-Evaluable Group |
| 14.2.3-7 | Specificity and Sensitivity of the Prostate Gland for Cohort A- Evaluable Set |
| 14.2.3-8 | Shift in Change of Management Questionnaire- Safety Set |
| 14.2.3-9 | Analysis of Change in Management Questionnaire- Safety Set |
| 14.2.3-10 | PPV and Positive Imaging from any tissue compared to histology for both Cohorts<br>Combined -Change in Management Set |
| 14.2.3-11 | Summary of Imaging Results-Safety Set |
| 14.2.3-12 | Summary of Histology Results- Safety Set |
| 14.2.3-13 | Summary of Procedures- Safety Set |
| 14.2.3-14 | Inter-Reader and Intra-Reader Variability for Cohort A- Evaluable Set |
| 14.2.4: Ef | 14.2.4: Efficacy- Per Protocol Set |
| 14.2.4-1 | Specificity and Sensitivity of the Pelvic Lymph Nodes for the Subjects in Cohort A- Per-Protocol Set |
| 14.3.1: Ad | lverse Events- Safety Set |
| 14.3.1-1 | Summary of Treatment Emergent Adverse Events, Overall and by Cohort -Safety Set |
| 14.3.1-2 | Most Frequent (>5% Overall) Treatment Emergent Adverse Events, Overall and by Cohort-Safety Set |
| 14.3.1-3 | Treatment Emergent Adverse Events Overall and by Cohort- Safety Set |
| 14.3.1-4 | Serious Treatment Emergent Adverse Events Overall and by Cohort- Safety Set |
| 14.3.1-5 | Drug Related Treatment Emergent Adverse Events Overall and by Cohort- Safety Set |
| 14.3.1-6 | Treatment Emergent Adverse Events where Severity Grade>=3, Overall and by Cohort-Safety Set |
| 14.3.1-7 | Treatment Emergent Adverse Events by Severity Grade, Overall – Safety Set |

| 14.3.2: Lis | sting of Deaths and Other Serious and Significant Adverse Events- Safety Set |
|---|---|
| 14.3.1-1 | Listing of Treatment Emergent Adverse Event Leading to Discontinuation or Death- Safety Set |
| 14.3.1-2 | Listing of Treatment Emergent Adverse Events Deemed Serious or With a Grade 3 or Above- Safety Set |
| 14.3.4: Ab | onormal Laboratory Value Listing |
| 14.3.4-1 | Listing of Abnormal Hematology Results – Safety Set |
| 14.3.4-2 | Listing of Abnormal Chemistry Results- Safety Set |
| 14.3.5: Vi | tal Signs |
| 14.3.5-1 | Summary and Change from Baseline in Vital Signs- Safety Set |
| 14.3.6: Ot | her Safety Data |
| 14.3.6-1 | Summary and Change from Baseline in Hematology Results- Safety Set |
| 14.3.6-2 | Summary and Change from Baseline in Chemistry Results- Safety Set |
| 14.3.6-3 | Clinical Laboratory Shift Table: Chemistry- Safety Set |
| 14.3.6-4 | Clinical Laboratory Shift Table: Hematology- Safety Set |
| 14.3.6-5 | Summary and Change from Baseline in ECG Parameters- Safety Set |
| 14.3.6-6 | Concomitant Medications- Safety Set |
| 14.3.6-7 | Study Drug Exposure- Safety Set |
| 14.4: PK I | Evaluations |
| 14.4-1 | Percent of Dose Recovered in Urine per Collection Interval -PK Urine Set |
| 14.4-2 | Summary of Urinary Kinetics- PK Urine Set |
| Listings | |
| 16.2.1-1 | Listing of Discontinuations – Consented Population |
| 16.2.2-1 | Listing of Protocol Deviations – Safety Set |
| 16.2.3-1 | Listing of Subjects Excluded from the Evaluable Set Used for Efficacy- Safety Set |
| 16.2.4-1 | Listing of Demographics- Consented Set |
| 16.2.5-1 | Listing of Blood PK by Nominal Blood Draw Times – PK Blood Set |
| 16.2.5-2 | Listing of Plasma PK by Nominal Blood Draw Times- PK Blood Set |
| 16.2.5-3 | Listing of Blood PK Parameters- PK Blood Set |
| 16.2.5-4 | Listing of Urinary Kinetics- PK Urine Set |
| 16.2.5-5 | Listing of Urine PK by Collection Intervals- PK Urine Set |
| 16.2.5-6 | Listing of Decay Corrected Dose – Safety Set |
| 16.2.5-7 | Listing of Compliance- Safety Set |
| 16.2.6-1 | Listing of Diagnostic Performance – Evaluable Set |

## Progenics Pharmaceuticals, Inc. Statistical Analysis Plan – Protocol PyL-2301

September 5, 2018

| 16.2.7-1 | Listing of Adverse Events- Safety Population |
|----------|----------------------------------------------|
| 16.2.8-1 | Listing of Laboratory Parameters- Safety Set |
| Figures | |
| riguies | |